CLINICAL TRIAL: NCT07274566
Title: The Effects of an 8-Week Exer-Genie-Assisted Speed and ABC Drill Training Program on Speed, Hamstring Strength, and Vertical Jump Performance in Female Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Rumeli University (Other)
Responsible Party: Principal Investigator, Yusufcan Keskin, PhD Student / Research Assistant, Istanbul Gedik University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EXERGENIE-FOOTBALL-2025
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Athletic Performance; Muscle Strength; Hamstring Muscles
Keywords: Resistance Training; Athletic Performance; Football

STUDY DESIGN:
Intervention Model Description: "Participants are randomly assigned to either the experimental group (Exer-Genie training) or the control group (standard training)."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in this group performed an Exer-Genie®-assisted sprint and agility-balance-coordination (ABC drill) training program twice per week for eight weeks in addition to their warm-up routine.
  Interventions: Other: Exer-Genie® Training Protocol
- Control Group (No Intervention): Participants in this group continued with their regular team football training only and did not receive the Exer-Genie® resistance training.

INTERVENTIONS:
Other: Exer-Genie® Training Protocol — The protocol consisted of six 30-m sprint runs performed with resistance applied using the 60-m Exer-Genie® device. Resistance was set at 10% of the athlete's body weight. The training was conducted twice a week for 8 weeks.
  Arms: Experimental Group

SUMMARY:
This study aims to examine the effects of an eight-week Exer-Genie®-assisted speed and agility-balance-coordination (ABC drill) training program on sprint performance, hamstring muscle strength, and vertical jump ability in young female football players. A total of 37 licensed female football players competing in the Turkish Women's Second League participated in the study. Participants were randomly assigned to an experimental group (n = 20) or a control group (n = 17). The study evaluates whether this integrated training approach enhances acceleration, force production, and neuromuscular control compared to regular team training alone.

DETAILED DESCRIPTION:
Study Design and Participants The study involves 37 female football players from the Pendik Güven Women's Football Team (mean age 14.4 ± 1.4 years), licensed by the Turkish Football Federation. Participants were randomly assigned to an experimental group (n = 20) or a control group (n = 17).

Intervention Protocol The experimental group completed an Exer-Genie®-assisted sprint and ABC drill training program twice per week for eight weeks (total of 16 sessions). Each session was performed after a standardized warm-up and consisted of six 30-m sprint runs and technical drills. The sprints were performed with resistance applied using the 60-m Exer-Genie® device, with resistance intensity set at 10% of each athlete's body weight. The control group continued with their regular team training only.Outcome Measures 1. Sprint Performance: Assessed via 0-10 m, 10-30 m, and 30 m sprint times using the SmartSpeed electronic timing gate system. 2. Hamstring Strength: Assessed using the NordBord Hamstring Testing System. Specifically, the ISO Prone (0°) protocol was used to measure isometric hamstring strength and impulse values. 3. Vertical Jump: Assessed via the Countermovement Jump (CMJ) test using the ForceDecks system to evaluate lower-limb explosive performance.Statistical Analysis Data were analyzed using repeated-measures ANOVA to evaluate time, group, and interaction effects, with a significance level set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Female gender.

Licensed football players competing in the Turkish Women's Second League.

Regularly engaged in football training for at least two years.

Aged between 11 and 17 years.

Exclusion Criteria:

History of recent musculoskeletal injury.

Any chronic health condition that could affect athletic performance.

Irregular attendance to the training sessions during the study period.

Ages: 11 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Sprint Performance (30m Sprint Test) | Baseline (Pre-test) and immediately after the 8-week intervention (Post-test)
  Sprint performance was evaluated using the SmartSpeed electronic timing gate system. Time was recorded in seconds for 0-10 m (acceleration), 10-30 m (transition), and full 30 m distances. Lower time indicates better performance.
Hamstring Muscle Strength (NordBord ISO Prone) | Baseline (Pre-test) and immediately after the 8-week intervention (Post-test)
  Isometric hamstring strength and impulse (force-time curve area) were assessed using the NordBord Hamstring Testing System with the ISO Prone protocol (0 degrees knee extension). Measured in Newtons (N) and N.s.
Vertical Jump Height (Countermovement Jump) | Baseline (Pre-test) and immediately after the 8-week intervention (Post-test)
  Lower-limb explosive power was assessed via the Countermovement Jump (CMJ) test using ForceDecks force platforms. Jump height was recorded in centimeters (cm).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Gedik University, Faculty of Sport Sciences, Indoor Sports Hall, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
"The datasets generated and analyzed during the current study are available from the corresponding author on reasonable request."
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning immediately after publication of the study results.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Requests should be directed to the corresponding author (Yusufcan Keskin) via email.